CLINICAL TRIAL: NCT04886622
Title: A Phase 1, Dose Escalation and Cohort Expansion Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of DT2216, an Antiapoptotic Protein Targeted Degradation Compound, in Patients With Relapsed/Refractory Malignancies
Brief Title: A Study of DT2216 in Relapsed/Refractory Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dialectic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DT2216-001
Record Dates: First submitted 2021-04-29; First posted 2021-05-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — DT2216

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DT2216 (Experimental): DT2216 will be administered by intravenous infusion over 30 minutes twice weekly on a continuous basis. Each treatment cycle will be 28 days in duration. The starting dose of DT2216 will be 0.04 mg/kg and will escalate by 100% increments for the first 5 treatment groups. Thereafter, if additional dose escalations are required, escalation will follow a modified Fibonacci scheme. Treatment may continue for up to 1 year.
  Interventions: Drug: DT2216

INTERVENTIONS:
Drug: DT2216 — DT2216 will be administered by intravenous infusion

SUMMARY:
A Phase 1, Open-Label, Dose Escalation, and Cohort Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Clinical Activity of DT2216, an Antiapoptotic Protein Targeted Degradation Compound, in Subjects with Relapsed or Refractory Malignancies

DETAILED DESCRIPTION:
This study is an open-label, first-in-human, dose escalation study in subjects with histologically or cytologically confirmed advanced or metastatic malignancies who are no longer responsive to approved or accepted standard-of-care interventions. The study will consist of a dose escalation phase followed by confirmation of the recommended phase 2 dose (RP2D).

Potentially eligible subjects will undergo screening evaluations (up to 28 days prior to study therapy) and those who meet all protocol-defined eligibility criteria will be enrolled into the study. Subjects who fail screening may be re-screened one time following correction or mitigation of the condition that caused the screen failure; there is no time limit on when a subject may be re-screened. Enrolled subjects will receive a single intravenous (IV) infusion of study drug on Days 1 and 4 weekly for at least 4 weeks, with each cycle consisting of 28 days. Treatment duration for an individual subject may continue for a maximum of 1 year, until disease progression, unacceptable toxicity, subject withdrawal, Investigator's decision for a change in treatment strategy for the individual subject, or death. Longer therapy may be considered for individual subjects upon consultation with the Sponsor's Medical Monitor and overall assessment of benefit:risk. Subjects will be followed for safety for 28 days following the administration of the last study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older on the day of signing informed consent.
2. Provide written informed consent for the trial, including willingness to comply with all study related requirements.
3. Histologically or cytologically confirmed solid tumor. Subjects with more than 1 primary malignancy may be considered upon review with the Sponsor's Medical Monitor
4. Evidence of disease progression or inadequate response on the last regimen as assessed by the Investigator.
5. Has exhausted all curative options or has a contraindication to approved therapies or generally recognized standard-of-care measures for the subject's cancer.
6. Presence of measurable disease as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
7. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Has adequate organ functions as defined by the following laboratory parameters at baseline (laboratory parameters outside of these ranges that are deemed clinically insignificant should be discussed with the Medical Monitor): (a) Absolute neutrophil count ≥1.5 x 109/L; (b) hemoglobin ≥9 g/dL; (c) platelet count ≥100,000/mm3; (d) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN); (e) total bilirubin ≤ 1.5 x institutional ULN (exception: subjects with known Gilbert's syndrome and total bilirubin ≤3.0 x ULN at screening or anytime during the prior 6 months are eligible); (f) c) adequate renal function defined as calculated creatinine clearance >60 mL/min using the Cockcroft-Gault Method (Appendix 3); (g) acceptable coagulation parameters including international normalized ratio (INR) <1.5 and partial thromboplastin time (PTT) ≤ institutional ULN; (h) serum albumin ≥3.0 g/dL.
9. Left ventricular ejection fraction of ≥50% as assessed by echocardiogram or multi-gated acquisition (MUGA) scan.
10. Adequate washout from the following prior to first dose of study therapy: Palliative radiation ≥ 2 weeks; chemotherapy or targeted therapy ≥ 3 weeks or 5 half-lives; biologic therapy ≥ 4 weeks.
11. Resolution to Grade ≤1 by the National Cancer Institute CTCAE, Version 5.0 (NCI-CTCAE v 5.0) of all clinically significant toxic effects of prior therapies.
12. Female subjects: A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: (a) Not a woman of childbearing potential (WOCBP); (b) WOCBP who agrees to follow the contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.
13. Female subject of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving any dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Male subject is eligible to participate if he agrees to follow the acceptable contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.

    -

Exclusion Criteria:

Diagnosis and Main Criteria for Inclusion:

Subjects are eligible to be included in the study only if all of the following criteria are met:

Inclusion Criteria

1. Adults aged 18 years or older on the day of signing informed consent.
2. Provide written informed consent for the trial, including willingness to comply with all study related requirements.
3. Histologically or cytologically confirmed solid tumor. Subjects with more than 1 primary malignancy may be considered upon review with the Sponsor's Medical Monitor.
4. Evidence of disease progression or inadequate response on the last regimen as assessed by the Investigator.
5. Has exhausted all curative options or has a contraindication to approved therapies or generally recognized standard-of-care measures for the subject's cancer.
6. Presence of measurable disease as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
7. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Has adequate organ functions as defined by the following laboratory parameters at baseline (laboratory parameters outside of these ranges that are deemed clinically insignificant should be discussed with the Medical Monitor): (a) Absolute neutrophil count ≥1.5 x 109/L; (b) hemoglobin ≥9 g/dL; (c) platelet count ≥100,000/mm3; (d) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN); (e) total bilirubin ≤ 1.5 x institutional ULN (exception: subjects with known Gilbert's syndrome and total bilirubin ≤3.0 x ULN at screening or anytime during the prior 6 months are eligible); (f) c) adequate renal function defined as calculated creatinine clearance >60 mL/min using the Cockcroft-Gault Method (Appendix 3); (g) acceptable coagulation parameters including international normalized ratio (INR) <1.5 and partial thromboplastin time (PTT) ≤ institutional ULN; (h) serum albumin ≥3.0 g/dL.
9. Left ventricular ejection fraction of ≥50% as assessed by echocardiogram or MUGA scan.
10. Adequate washout from the following prior to first dose of study therapy: Palliative radiation ≥ 2 weeks; chemotherapy or targeted therapy ≥ 3 weeks or 5 half-lives; biologic therapy ≥ 4 weeks.
11. Resolution to Grade ≤1 by the National Cancer Institute CTCAE, Version 5.0 (NCI-CTCAE v 5.0) of all clinically significant toxic effects of prior therapies.
12. Female subjects: A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: (a) Not a woman of childbearing potential (WOCBP); (b) WOCBP who agrees to follow the contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.
13. Female subject of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving any dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Male subject is eligible to participate if he agrees to follow the acceptable contraceptive guidance during the study treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria

1. Received any BCL-XL directed therapy.
2. Administration of any blood products within the 30 days preceding the planned administration of study therapy.
3. History of clinically significant bleeding and/or bleeding predisposition.
4. Significant liver insufficiency defined as Child-Pugh Class B or C
5. Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A (CYP3A). Strong CYP3A inhibitors and inducers should be discontinued at least 2 weeks prior to the first dose of DT2216 (Appendix 5).
6. Known active central nervous system (CNS) metastases/and or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable without evidence of progression via imaging for at least 4 weeks prior to first dose of study therapy, are not receiving pharmacologic doses of glucocorticoids and are without evidence of neurological symptoms. Carcinomatous meningitis is excluded regardless of clinical stability.
7. Requiring anticoagulation for any reason (subjects who are on anticoagulants during the screening period and are candidates for discontinuation can be considered).
8. Prior organ transplantation including allogeneic or autologous stem-cell transplantation or other cellular therapies (e.g. chimeric antigen receptor T-cells [CAR-T]).
9. Major surgery <4 weeks prior to first dose of study therapy.
10. Growth factor use <4 weeks prior to first dose of study therapy.
11. Participation in another research study involving receipt of an investigational product <4 weeks prior to first dose of study therapy. If the half-life of the investigational study is known, a shorter interval may be appropriate and should be discussed with the Sponsor's Medical Monitor. Participants who have entered the follow-up phase of an investigational study may be eligible as long as it has been 4 weeks after the last dose of the previous investigational agent.
12. Active autoimmune disease or history of chronic recurrent autoimmune disease, requiring systemic treatment for the past 2 years (i.e. disease modifying agents, corticosteroids or immunosuppressive drugs). Hormone replacement therapy (thyroxine, insulin, or physiological corticosteroid replacement for either adrenal or pituitary insufficiency) is not considered a form of systemic treatment directed at an autoimmune disorder.
13. Systemic steroid therapy (>10 mg daily prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment (note: topical, inhaled, nasal and ophthalmic steroids are permitted).
14. Known active hepatitis B (e.g, HBsAg reactive), hepatitis C (HCV) (e.g., HCV RNA [qualitative] is detected). Subjects who have completed a course of anti-viral therapy for hepatitis C and are polymerase chain reaction (PCR) negative are eligible.
15. Active infection with human immunodeficiency virus (HIV) unless: (a) Subject is currently off antiretroviral therapy (ART) for at least 4 weeks; (b) HIV viral load of < 400 copies per milliliter (/mL) at Screening (or undetectable per local criteria); (c) cluster of differentiation (CD4) counts ≥200/microliter
16. Active infection requiring systemic therapy.
17. Known allergy to any component of the study treatment formulation(s).
18. Known history of marked prolongation of the QT or QT corrected (QT /QTc) interval or a mean QTc as assessed by Fridericia's method (QTcF) value >470 msec following 3 ECG determinations 5 minutes apart at Screening.
19. History of additional risk factors for Torsade de Pointes (including heart failure, hypokalemia, family history of Long QT Syndrome, and use of concomitant medications that prolong the QT/QTc interval.
20. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of study treatment.
21. Clinically significant cardiovascular disease including: History of myocardial infarction within 6 months prior to day 1 of study therapy, symptomatic congestive heart failure (New York Heart Association Class II to IV), unstable angina, or serious cardiac arrhythmia requiring treatment, uncontrolled angina within 3 months of day 1 of study therapy, uncontrolled hypertension.
22. Corona Virus Disease (COVID-19) diagnosis within 3 months of first dose of study drug.
23. Any other history of clinically significant and ongoing chronic respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder or any other medical or psychiatric condition that in the opinion of the Investigator will significantly increase the safety risk for the subject or confound the interpretation of the study data.
24. History of alcohol or drug abuse within 6 months of first dose of study therapy or a social situation that would interfere with the subject's participation in the trial.
25. In the opinion of the Investigator, participant has rapidly progressing disease, OR has life expectancy <3 months.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The number of subjects with adverse events based on the Common Terminology Criteria for Adverse Evens (CTCAE) v5.0 following treatment with DT2216. | 28 days
  The incidence of adverse events will be the number of subjects with an adverse event divided by the total number subjects.
The number of subjects with adverse events of different grades based on the CTCAE v5.0 | 28 days
  The severity will be based on the grading of adverse events as described in the CTCAE v5.0
The number of subjects with dose limiting toxicity (DLT) of DT2216. | 28 days
  DLT's will be defined by any of the following:
  Any Grade 5 toxicity on the CTCAE CTCAE v5.0 Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with clinically significant hemorrhage CTCAE Grade 4 neutropenia lasting >7 days Febrile Neutropenia, defined as absolute neutrophil count (ANC) <1000/mm3 with a single temperature of >38.3°C (101°F) or a sustained temperature of >38°C (100.4°F) for >1 hour Grade 3 thrombocytopenia that is clinically uncomplicated and lasting ≥7 days. CTCAE Grade 4 non-hematologic toxicity of any duration CTCAE Grade 3 non-hematologic toxicity, except nausea, vomiting and/or diarrhea lasting ≤3 days or laboratory abnormalities that return to baseline within ≤3 days with or without medical intervention Changes in liver enzymes consistent with Hy's law indicative of drug-induced hepatocellular injury

SECONDARY OUTCOMES:
The measurement of Cmax of DT2216 following intravenous administration | 28 days
  The Cmax will be based on blood levels following intravenous administrration of DT2216.
The measurement of the half-life of DT2216 following intravenous administartion | 28 days
  The half-life will be based on blood levels of DT2216 following intravenous administration.
The measurement of the clearance of DT2216 following intravenous administration. | 28 days
  The clearance of DT2216 will be based on blood levels of DT2216 following intravenous administration
The measurement of levels of BCL-XL in peripheral blood mononuclear cells | 28 days
  Levels of BCL-XL will be measured in peripheral blood mononuclear cells
The measurement of platelet counts following administration of DT2216 | 28 days
  Platelet counts will be determined at various time points after administration of DT2216
The number of subjects who have oncological responses to DT2216 based on the RECIST 1.1 criteria. | One year
  The response rate to DT2216 will be determined at various time points following administration of DT2216 based on the Response Evaluation Criteria in Solid Tumors 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Dialectic Therapeutics
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Mary Crowley Cancer Research, Dallas, Texas
  - Mays Cancer Center, San Antonio, Texas

REFERENCES:
- [Background] Khan S, Zhang X, Lv D, Zhang Q, He Y, Zhang P, Liu X, Thummuri D, Yuan Y, Wiegand JS, Pei J, Zhang W, Sharma A, McCurdy CR, Kuruvilla VM, Baran N, Ferrando AA, Kim YM, Rogojina A, Houghton PJ, Huang G, Hromas R, Konopleva M, Zheng G, Zhou D. A selective BCL-XL PROTAC degrader achieves safe and potent antitumor activity. Nat Med. 2019 Dec;25(12):1938-1947. doi: 10.1038/s41591-019-0668-z. Epub 2019 Dec 2. PMID 31792461
- [Derived] Mahadevan D, Barve M, Mahalingam D, Parekh J, Kurman M, Strauss J, Tremaine L, Hromas R, Sills J, McCulloch J, Harkey J, Suberg S, Zimmerman L, Zheng G, Zhou D. First in human phase 1 study of DT2216, a selective BCL-xL degrader, in patients with relapsed/refractory solid malignancies. J Hematol Oncol. 2025 Nov 12;18(1):98. doi: 10.1186/s13045-025-01753-8. PMID 41225624